CLINICAL TRIAL: NCT00451841
Title: Exhaled Breath Condensate pH in Patients With Cough Caused by Gastroesophageal Reflux
Status: Terminated | Type: Observational
Why Stopped: IRB approval not renewed/approval lapsed. Prior status: insufficient enrollment; study suspended pending analysis
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Stephen Krinzman, Principal Investigator, University of Massachusetts, Worcester
Other Study IDs: H-12073
Record Dates: First submitted 2007-03-22; First posted 2007-03-26 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Cough; Gastroesophageal Reflux
Keywords: Cough; Gastroesophageal reflux; Exhaled breath condensate
MeSH Terms: conditions — Cough; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — frozen sputum supernatant and exhaled breath condensate fixed sputum cell preparations
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Chronic cough caused by GERD
  Interventions: Device: RTube Exhaled Breath Condensate Collection System
- 2: Chronic cough without GERD
  Interventions: Device: RTube Exhaled Breath Condensate Collection System

INTERVENTIONS:
Device: RTube Exhaled Breath Condensate Collection System — Subjects breath through the device to collect exhaled breath condensate

SUMMARY:
Cough is the most common complaint for which patients seek medical attention in the United States, accounting for approximately 1 billion dollars in health care expenses annually. Gastroesophageal reflux disease (GERD) is the sole cause of chronic cough in up to 20-40% of all cases. The majority of these patients with GERD-induced cough have no classic "heartburn" symptoms, so this important cause of cough can thus be difficult to detect.

Our hypothesis is that changes in exhaled breath condensate (EBC) pH can be used as a sensitive and non-invasive marker to identify subjects with cough caused by acid reflux.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is the sole cause of chronic cough in up to 20-40% of all cases, and majority of these patients with GERD-induced cough have no classic "heartburn" symptoms. This important cause of cough can thus be difficult to detect. Non-invasive radiologic tests for GERD such as barium swallow is imperfectly sensitive in subjects with GERD-induced cough. The 24 hour pH probe, which continuously monitors esophageal pH and can correlate cough events with reflux events, is considered to be the gold standard test. However, this test is expensive, invasive, and not universally available.

The goal of the current study is to compare simultaneous measurements of esophageal pH with exhaled breath condensate pH after cough episodes, in patients with symptomatic cough. The cause of cough will be determined by a standard protocol, which includes 24 hour pH probe studies, and assessment for asthma, upper airway causes and sinus disease, and medication effects. All subjects will undergo 24 hour pH monitoring. During this monitoring period, they press an event button on the pH recording device to indicate a cough episode. After six such events, they will immediately perform an EBC collection, and EBC pH will subsequently be analyzed. Differences between pH changes in the group with cough cause by GERD will be compared to pH measurements in the group with cough but no GERD, to determine the sensitivity and specificity of pH changes for discriminating between the two groups, and optimal threshold values for pH changes in EBC.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* able to speak and read English
* chronic cough

Exclusion Criteria:

* Cigarette smoking within the past 6 months, or greater than 10 pack year history of prior smoking
* Any self-reported or clinically diagnosed form of active lung disease, including asthma and emphysema
* Symptoms of persistent rhinitis within the past three months
* Dysphagia
* Symptoms of acute viral upper respiratory tract infection or sinusitis within one month of entry into the study
* Pregnancy - based on self report
* Abnormal chest radiograph

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients evaluated for cough in the Lung and Allergy Center of Umass Memorial Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2007-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity of esophageal PH changes | 24 hours
  Determine the sensitivity of esophageal PH changes between the group with GERD and the group without GERD.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Krinzman, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- UMass Memorial Medical Center, University Campus, Worcester, Massachusetts, United States

REFERENCES:
- [Background] Niimi A, Nguyen LT, Usmani O, Mann B, Chung KF. Reduced pH and chloride levels in exhaled breath condensate of patients with chronic cough. Thorax. 2004 Jul;59(7):608-12. doi: 10.1136/thx.2003.012906. PMID 15223872
- [Background] Hunt J. Exhaled breath condensate pH: reflecting acidification of the airway at all levels. Am J Respir Crit Care Med. 2006 Feb 15;173(4):366-7. doi: 10.1164/rccm.2512001. No abstract available. PMID 16467175
- [Background] Horvath I, Hunt J, Barnes PJ, Alving K, Antczak A, Baraldi E, Becher G, van Beurden WJ, Corradi M, Dekhuijzen R, Dweik RA, Dwyer T, Effros R, Erzurum S, Gaston B, Gessner C, Greening A, Ho LP, Hohlfeld J, Jobsis Q, Laskowski D, Loukides S, Marlin D, Montuschi P, Olin AC, Redington AE, Reinhold P, van Rensen EL, Rubinstein I, Silkoff P, Toren K, Vass G, Vogelberg C, Wirtz H; ATS/ERS Task Force on Exhaled Breath Condensate. Exhaled breath condensate: methodological recommendations and unresolved questions. Eur Respir J. 2005 Sep;26(3):523-48. doi: 10.1183/09031936.05.00029705. PMID 16135737